CLINICAL TRIAL: NCT03122145
Title: Establishing Normal Swallowing and Breathing Profiles in Healthy Adults Across the Age Span
Brief Title: Normal Breathing and Swallowing in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201700132 - A
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: healthy; volunteer
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers - Experiment 1 (Experimental): This study will involve a single 60-minute visit. All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process during to radiation exposure. Eligible participants will then undergo voluntary and reflexive cough testing. The entire duration of the exam will be under 60 minutes and the participant will be free to leave at any point during the examination.
  Interventions: Drug: Capsaicin; Device: Videofluoroscopic swallow study
- Healthy Volunteers - Experiment 2 (Experimental): This study will involve a single 60-minute visit. All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process during to radiation exposure. Eligible participants will then undergo a instrumental swallowing evaluation (videofluoroscopy). The entire duration of the exam will be under 60 minutes and the participant will be free to leave at any point during the examination.
  Interventions: Device: Videofluoroscopic swallow study

INTERVENTIONS:
Drug: Capsaicin — Participants will inspire deeply through the nebulizer coupled to the facemask and pneumotachograph. Each test inhalation will be separated by an interval of 2 minutes. This experimental trial consists of six (instead of 8) test solutions: 0, 25, 50, 100, 200 and 500 μM capsaicin in 80% physiological saline, 20% ethanol. Participants will inhale single vital capacity breaths of capsaicin solution via an air-powered dosimeter (KoKoDigidoser; Pulmonary Data Services Instrumentation Inc; Louisville, CO). The reflex cough test ends when the participant coughs at least 2 times in response to one inhalation dose, or receives a dose of the highest concentration (500 μM).
  Other Names: Reflexive Cough
  Arms: Healthy Volunteers - Experiment 1
Device: Videofluoroscopic swallow study — The swallowing systems core laboratory is fully equipped to perform videofluoroscopy with a c-arm (OEC 9900) that is dedicated solely to research purposes. Videofluoroscopy recordings will be kept to a minimum and turned on only during completion of a specific testing task. Video recording and images captured during the videofluoroscopy will be synced and saved for data analysis. Videofluoroscopy allows for time-synced, frame-by-frame data analysis for the specific measures taken during swallowing tasks. The physiological swallowing measures (temporal and kinematic of the base of tongue, oropharynx, and hyolarynx complex during swallowing) to be analyzed cannot be visualized with any other technique. All swallowing tasks will be completed using barium in order to visualize the bolus during movement of various swallowing muscles and structures.

SUMMARY:
The purpose of this study is to establish normative values for clinical testing measures of swallow, respiratory and cough functions. This will aide in establishing degree of impairment in disordered populations, and in identifying efficacious treatment paradigms for dysphagia.

DETAILED DESCRIPTION:
The prevalence of dysphagia may be as high as 22% in individuals over 50 years of age. There are few therapeutic options and minimal management strategies offered to treat these individuals and improve sequelae of dysphagia. Dysphagia contributes to malnutrition, aspiration, pneumonia, reduced quality of life and increased mortality in neurodegenerative disease such as ALS. One reason for this is the lack of normative data across various measures of swallowing and respiratory function. As a result, detecting early impairments in swallowing physiology is difficult, given the variability of swallowing and unknown normative value range of swallowing physiology. Therefore, the goal of this study is to complete clinical tests of swallowing and cough function in healthy volunteers to establish normative data. This will contribute to future study in disordered populations, to determine degree and severity of impairment and efficacious treatment and management strategies based on impairment.

The purpose of this study is to establish normative values for clinical testing measures of swallow, respiratory and cough functions. This will aide in establishing degree of impairment in disordered populations, and in identifying efficacious treatment paradigms for dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Up to 120 individuals will be included in this study.
* Subjects will include both male and females who are aged between 18-100
* Healthy and with no major medical conditions.
* No specific gender or race will be excluded or targeted for participation in this study.

Exclusion Criteria:

* Adults who are pregnant
* Those with major medical conditions (i.e., swallowing impairment, brain injury) will be excluded from this study.
* Anyone with allergy to barium will be excluded from this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The study team will not be sharing individual IDP information with other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2018-2019 HealthStreet university approved flyers
Pre-assignment Details: Experiment #1: single 60 minute visit with multiple assessments of cough and respiratory function.
  Experiment #2: single 60-minute visit with an instrumental swallowing evaluation (videofluoroscopy).
Groups:
- Healthy Volunteers - Experiment #1: This study will involve a single 60-minute visit where healthy, eligible participants will then undergo testing to determine their individualized voluntary and reflexive cough testing. The participant will be free to leave at any point during the examination.
  Capsaicin: Participants will inspire deeply through the nebulizer coupled to the facemask and pneumotachograph. Each test inhalation will be separated by an interval of 2 minutes. This experimental trial consists of six test solutions: 0, 25, 50, 100, 200 and 500 μM capsaicin in 80% physiological saline, 20% ethanol. Participants will inhale single vital capacity breaths of capsaicin solution via an air-powered dosimeter (KoKoDigidoser).
- Healthy Volunteers - Experiment #2: This study will involve a single 60-minute visit eligible participants will then undergo an instrumental swallowing evaluation (videofluoroscopy). All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process prior to radiation exposure. The entire duration of the exam will be under 60 minutes and the participant will be free to leave at any point during the examination.
Period: Overall Study
Arm/Group | Healthy Volunteers - Experiment #1 | Healthy Volunteers - Experiment #2
Started | 37 (34 participants completed the first sub study under this IRB) | 12
Completed | 34 | 12
Not Completed | 3 | 0
Not completed — Concurrent respiratory disease | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants were healthy controls recruited from the Gainesville community and university population.
Groups:
- Healthy Volunteers - Experiment #1: This study will involve a single 60-minute visit where healthy, eligible participants will undergo testing to determine their individualized voluntary and reflexive cough testing. The participant will be free to leave at any point during the examination.
- Healthy Volunteers - Experiment #2: This study will involve a single 60-minute visit where healthy, eligible participants will undergo an instrumental swallowing evaluation (videofluoroscopy). All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process during to radiation exposure. The participant will be free to leave at any point during the examination.
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers - Experiment #1 | Healthy Volunteers - Experiment #2 | Total
Number analyzed (Participants) | 34 | 12 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 12 | 30
  >=65 years | 16 | 0 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (15.22) | 27 (3.86) | 52 (18.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 14 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 25 | 0 | 25
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 2 | 12 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 12 | 46

OUTCOME MEASURES:

1. Primary Outcome: Reflexive Cough Testing (With Urge-to-Cough)
Description: Reflexive cough testing will use a capsaicin challenge that will assess individual's cough motor and cough sensory thresholds. A modified Borg scale ranging from 0 (no cough) to 10 (maximal urge to cough) will be used to quantify these thresholds. A cough sensory threshold will be defined as a concentration of capsaicin eliciting a perceived urge to cough of 1 (very slight) >2/3 trials. A cough motor threshold will be the lowest concentration of capsaicin eliciting >2 cough responses in 2/3 trials.
Time Frame: Single assessment time period
Population: Participants who completed the entire randomized reflex cough testing protocol were included in the analysis
Measure: Median (Full Range); unit: units on a scale
Groups:
- Healthy Volunteers: This study will involve a single 90-minute visit. All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process during to radiation exposure. Eligible participants will then undergo voluntary and reflexive cough testing, tongue pressure testing and a comprehensive instrumental swallowing evaluation. The entire duration of the exam will be under 90 minutes and the participant will be free to leave at any point during the examination.
  Capsaicin: Participants will inspire deeply through the nebulizer coupled to the facemask and pneumotachograph. Each test inhalation will be separated by an interval of 2 minutes. This experimental trial consists of six (instead of 8) test solutions: 0, 25, 50, 100, 200 and 500 μM capsaicin in
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 34
units on a scale
  cough motor threshold | 3 [0 to 10]
  cough sensory threshold | 5 [0.5 to 10]

2. Primary Outcome: Duration of Laryngeal Vestibule Closure (dLVC)
Description: LVC temporal measures will be used to calculate the duration of laryngeal vestibule closure (dLVC)
Time Frame: Single Visit
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- Healthy Volunteers - Experiment 2: This study will involve a single 60-minute visit. All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process during to radiation exposure. Eligible participants will then undergo a instrumental swallowing evaluation (videofluoroscopy). The entire duration of the exam will be under 60 minutes and the participant will be free to leave at any point during the examination.
  Videofluoroscopic swallow study: The swallowing systems core laboratory is fully equipped to perform videofluoroscopy with a c-arm (OEC 9900) that is dedicated solely to research purposes. Videofluoroscopy recordings will be kept to a minimum and turned on only during completion of a specific testing task. Video recording and images captured during the videofluoroscopy will be synced and saved for data analysis. Videofluoroscopy allows for time-synced, frame-by-frame data analysis for the specific measures taken during swallowing tasks.
Arm/Group | Healthy Volunteers - Experiment 2
Number analyzed (Participants) | 12
Milliseconds
  5 swallows with head in chin up position | 435 (41)
  5 swallows with e-stim to anterior neck | 429 (61)
  5 swallows with head in neutral position | 461 (39)

3. Secondary Outcome: Voluntary Peak Cough Flow Testing (With Electronic Peak Cough Flow Meter Device)
Description: Voluntary peak cough flow testing will be used to capture the volume of air expelled in the 1st second of cough as measured in PEF and FEV1.
Time Frame: Baseline
Population: Participants who completed the voluntary cough testing protocol in its entirety were included in the analysis
Measure: Mean (Standard Deviation); unit: liters per second
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 34
liters per second | 3.15 (1.01)
Statistical Analysis 1: Comparison: Healthy Volunteers; Hypothesis that voluntary cough > reflex cough strength and effectiveness in healthy volunteers; Test type: Superiority — Mann whitney U between groups comparison for voluntary cough parameters between healthy controls and individuals with ALS outcomes: peak expiratory cough flow and cough volume acceleration; p = 0.0005, ANOVA

4. Primary Outcome: Laryngeal Vestibule Closure Reaction Time (LVCrt)
Description: LVC temporal measures will be used to calculate the laryngeal vestibule closure reaction time (LVCrt)
Time Frame: Single Visit
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Healthy Volunteers - Experiment 2
Number analyzed (Participants) | 12
Milliseconds
  5 swallows with head in chin up position | 181 (31)
  5 swallows with e-stim to anterior neck | 174 (23)
  5 swallows with head in neutral position | 169 (34)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Other (adverse event reporting): adverse events related to voluntary and reflex cough testing were collected during the single testing session. Participants were briefly monitored after testing and study was completed following their single visit.
Groups:
- Healthy Volunteers - Experiment #1: This study will involve a single 60-minute visit where healthy, eligible participants will undergo voluntary and reflexive cough testing.
  Capsaicin: Participants will inspire deeply through the nebulizer coupled to the facemask and pneumotachograph. Each test inhalation will be separated by an interval of 2 minutes. This experimental trial consists of six (instead of 8) test solutions: 0, 25, 50, 100, 200 and 500 μM capsaicin
- Healthy Volunteers - Experiment #2: This study will involve a single 60-minute visit where eligible participants will undergo an instrumental swallowing evaluation (videofluoroscopy). All women under the age of 62 will be asked to complete a pregnancy test as part of the screening process prior to radiation exposure. The entire duration of the exam will be under 60 minutes and the participant will be free to leave at any point during the examination.
Arm/Group | Healthy Volunteers - Experiment #1 | Healthy Volunteers - Experiment #2
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/12
Other Adverse Events (participants affected / at risk) | 1/34 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers - Experiment #1 (N=34) | Healthy Volunteers - Experiment #2 (N=12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Reported shortness of breath following the maximum capsaicin dose during reflex cough testing. Participant was provided water and took a 5-minute break. They completed the study without issue and were sent home after a brief monitoring period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03122145/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03122145/SAP_001.pdf